CLINICAL TRIAL: NCT05648617
Title: Effectiveness of Protein Supplementation on Frailty Improvement, Muscle Strength and Physical Performance Among Pre-Frail Elderly People in Selangor- Malaysia: A Randomized Clinical Study
Brief Title: Effectiveness of Protein Supplementation on Frailty Improvement, Muscle Strength and Physical Performance Among Pre-Frail Elderly People
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Alaa Hussein Alrawhani, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UPM UNIVERSITY
Record Dates: First submitted 2022-11-12; First posted 2022-12-13 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Frailty; Muscle Weakness; Physical Dependence; Weight Loss
Keywords: Frailty; Protein Supplements; Elderlies; Muscle Strength; Physical Performance
MeSH Terms: conditions — Frailty; Muscle Weakness; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Protein Supplement group (Active Comparator): Participants will receive 30g of SUSTINEX Hydrolyzed Whey Protein supplement. The participants will be asked to add it to their soft food or their beverages to reach the goal of consuming 30g daily for 12 weeks (3months).
  Interventions: Dietary Supplement: SUSTINEX Hydrolyzed Whey Protein
- control group (No Intervention): Receive no intervention- usual care, will receive the standard care of the clinic without supplemented with PS.

INTERVENTIONS:
Dietary Supplement: SUSTINEX Hydrolyzed Whey Protein — Participants will receive 30g of SUSTINEX Hydrolyzed Whey Protein. The participants will be asked to add it to = to reach the goal of consuming 30g daily. SUSTINEX Whey Protein Plus is an authorized protein supplement which is manufactured and made in Malaysia by Nova Laboratories Sdn. Bhd. (179832-D). It consists of whey protein isolate and whey protein hydrolyze to achieve sufficient protein requirement.
  Arms: Protein Supplement group

SUMMARY:
The goal of this randomized clinical trial is to study the effectiveness of protein supplements in frailty improvement, muscle strength, physical performance, energy intake and body composition of pre-frail elderly people. in Selangor, Malaysia.

The main question[s] it aims to answer are:

Does PS intervention significantly affect in frailty improvement, muscle strength, physical performance, energy intake and body composition of elderly people? For the interventional group, Participants will receive 30g of SUSTINEX Hydrolyzed Whey Protein. The participants will be asked to add it to their food or drinks to reach the goal of consuming 30g daily. For control group, participants will receive no intervention- usual care, will receive the standard care of the clinic without supplemented with PS.

DETAILED DESCRIPTION:
Several studies stated that an increase in dietary protein consumption may help to prevent muscle loss and stimulate muscle protein synthesis. This study aims to study the effectiveness of protein supplements in frailty improvement, muscle strength, physical performance, energy intake and body composition of pre-frail elderly people. This study is a 3-months (12 weeks), single blind, parallel randomized controlled experiment with two arms in which outpatient persons in Serdang hospitals, Malaysia, are randomly assigned to one of two arms: a) control group (CG), and b) protein (PSG) supplementation in two of Selangor hospital's outpatients (Serdang Hospital, Hospital Pengajar UPM) Serdang, Malaysia. Study population are men or women elderlies who 60 years or more and classified (according to Fried criteria) as pre-frail older adults.

Sample size was calculated based on the findings of (Shahar et al., 2019), considering a mean ± SD of BMI in protein supplement study as 25.91 ± 2.96 kg/m2 in the placebo group and 23.82 ± 4.16 kg in protein supplement group, with a power of 80% and an α level (2-tailed) of 5%. This process conducted using G Software. This gave a sample size of 17 participants/group and total 34 participants. With an expected dropout rate of 20%, a sample size of 20 participants/group is considered adequate.

* Participants will be recruited from outpatient and Dietetics clinics patients who will be screened by the site investigators in both Serdang and HPUPM hospital using FRAIL Screen and demographic and health-related information will be collected.
* An information papers will be given and discussed following the invitation procedure. Individuals who agree to participate will be asked to submit written informed permission and will then be screened to determine their eligibility to participate. Individuals who have been assessed as eligible to participate will be invited to a pre-intervention data collection session (baseline assessment).
* After testing the eligibility, a random sequence will be generated for the patients' numbers which results in a sequence of random numbers divided in two groups.
* The allocation ratio is 1:1. To guarantee allocation concealment, the randomization will be carried out by an independent third party. The envelope will be opened on the spot, deciding which group the participant would be allocated to either Group 1 (PSG): Intervention Group or Group 2 (CG): Control Group.

Protein Supplement Group:

Participants will receive 30g of SUSTINEX Hydrolysed Whey Protein. The participants will be asked to add it to their soft food or their beverages to reach the goal of consuming 30g daily.

Control Group (CG) Receive no intervention- usual care, will receive the standard care of the clinic without supplemented with PS.

• Before entering the run-in period, the participants will be interviewed using a structured questionnaire to obtain information: Demographic data of participants, anthropometric measurements, practice function/performance, muscle strength activities, dietary intake (3-day food record) will all be done one week prior to the intervention period in order to get the baseline data.

Interventional group:

* All participants will be instructed on how to prepare and consume the protein supplements and how to record them in the provided compliance diaries.
* The supplement will be in powder form in individual sachets (15g per sachet) and subjects will be asked to mix 2 sachets daily in their soft foods or beverages (1 sachet in the morning & 1 sachet in the evening).

Supplements Supplying:

• Supplements will be handed to the participants in the dietetic clinic at the beginning of the trial and in the middle (6th week) of the trial and they will be asked to return the previous can in order to check the retain sachets.

Monitoring Process:

* Compliance diaries will be handed out to participants with instructions provided on how to complete them; specifically, they will be asked to record the timing and number of supplements consumed per day.
* The researcher will check compliance with the supplements prescription on a weekly- basis message reminder sent to each participant.
* According to the remained sachets and the dairies, if the study team identify that a participant's compliance to the planned number of protein sachets, is less than 70%, the researcher will respectively interview the participant to assess any difficulties and identify strategies that could facilitate compliance.

Follow-up Process:

* Participants should not take any over-the-counter medications without informing the researcher. They can continue taking the prescribed medications by their respective physicians.
* Adverse events (AEs), that is, any untoward medical occurrences will be investigated during all visits, whether or not they are related to the study product. The events will be reviewed by the study's investigator and participants will be referred to the research physician as required.

Data analysis The research design is structured on two assessments which involves the baseline and after the intervention. The characteristics of the baseline respondents (CG, PSG) will be reported. Missing data at random (MAR) method will be used treat data that are missing during intervention by way of intention to treat (ITT) as recommended by Dziura, Post, Zhao, Fu, & Peduzzi (2013).

Categorical variables will be summarized by frequencies and percentages, continuous variables will be summarized by means and standard deviation. Additionally, cross tabulation of the categorical variables will be done to verify the independency of some required variables targeted in the research objectives which will be verify via chi-square test or Fisher's exact test.

The continuous data will further be examined for conformity to normality distribution assumptions, the continuous data with non-normality characteristics will be summarized by the median (IQR). Non-parametric statistical methodology such as Mann Whitney, Wilcoxon signed rank test among other statistical methodologies will be adopted accordingly for non normal continuous variables.

Analysis of variance (ANOVA) on repeated measures for the second factor will be used to assess variability in weight loss, exhaustion, weakness, slowness and low activity between the baseline and intervention. Analysis of covariance (ANCOVA) via generalized linear model will be adopted for the post-intervention analysis. The sensitivity analysis will be examined through receiver operating characteristics (ROC) curves especially on variables that has missing data.

ELIGIBILITY:
Inclusion Criteria:

* Pre-frail men or women aged 60 years and above (Fried criteria: score ≥1 but <3 out of 5).
* Willing to give informed consent to be randomized to either the protein supplement or control group
* Willing to follow the study protocol.

Exclusion Criteria:

* Non or Frail elderlies (Fried criteria)
* Diagnosed with chronic diseases include: (heart-related disease, COPD, stroke, cancer, asthma, renal dysfunction, terminally ill), bedridden.
* Already involved or still participating in any health interventional studies.
* Participants who consume protein supplements
* Any sustained fracture (hip, vertebrata) in past six month, any surgery (hip, abdominal area) in past six month

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
To study the differences in frailty status, scores and its phenotypes for protein supplemented group (PSG) and control group (CG) from pre- and post-intervention (3 months after intervention starts) in the prefrail elderlies. | Baseline & after 12 weeks of the intervention.
  To study the change of frailty phenotypes (Weight loss/ shrinking - Exhaustion - Weakness - Slowness - Low activity) will be measured according to Fried Criteria using report sheet ≥ 3 frailty Criteria = Frail
  1 - 2 frailty Criteria = Pre-frail 0 frailty Criteria = Normal.
To compare the changes in body weight, lean body mass, muscle mass, total body fat for protein supplemented group (PSG) and control group (CG) from pre- and post-intervention (3 months after intervention starts) in the prefrail elderlies. | Baseline, 6th, and 12th week of the intervention.
  Body weight, lean body mass, total body fat (TBF), and muscle mass will be measured to the nearest 0.1 kg using whole-body dual-energy X-ray absorptiometry DXA and a portable body composition analyzer (OMRON HBF-375, Japan).
To compare pre- and post-intervention changes in Body Mass Index BMI, for the interventional group (PSG) and control group (CG) in the prefrail elderly. | Baseline, 6th, and 12th week of the intervention.
  BMI will be calculated as the body mass in kilograms divided by the square of the height in meters. Standing height (±1.0 cm) will be measured using a wall stadiometer.
To assess pre- and post-intervention score changes in the balance test, one of the short physical performance battery (SPPB) tests, for the interventional group (PSG) and control group (CG) in the prefrail elderly. | Baseline, 6th, and 12th week of the intervention.
  Balance tests comprises the duration of each of side-by-side stand, semitandem stand, and tandem stand; the duration of each stand is 10 seconds, if the participant can hold this duration, 1 point will be awarded, except for the tandem stand, which is worth 2 points for this duration.
To compare pre- and post-intervention score changes in the gait speed test, one of the short physical performance battery (SPPB) tests, for the interventional group (PSG) and control group (CG) in the prefrail elderly. | Baseline, 6th, and 12th week of the intervention.
  The gait speed test is the time to complete a 4-meter walk (repeated 3 times); the score for this test is graded from 0 to 4; 0 means the participant was unable to do the walk, and 4 means the time taken to complete the 4-meter walk was less than 4.8 seconds.
To compare pre- and post-intervention score changes in the sit-to-stand test, the third component of the short physical performance battery (SPPB) tests, for the interventional group (PSG) and control group (CG) in the prefrail elderly. | Baseline, 6th, and 12th week of the intervention.
  The sit-to-stand test is the time to rise from sitting (repeated 5 times),the score will be graded from 0 to 4; 0 means the participant was unable to complete 5 chair stands or complete stands in more than 60 seconds, and 4 means the chair stand time is 11.19 seconds or less.
To assess pre- and post-intervention physical performance level changes using short physical performance battery (SPPB) tests, for the interventional group (PSG) and control group (CG) in the prefrail elderly. | Baseline, 6th, and 12th week of the intervention.
  The SPPB consists of balance, gait speed, and sit-to-stand ability. A 0- to 12-point scale is used to score the sum of the three assessments, with higher point values corresponding with greater levels of physical function and lower disability, whereas lower point values correspond with lower levels of physical function and higher disability, respectively.
To assess the changes in the muscle strength for interventional group (PSG) and control group (CG) from pre- and post-intervention (3 months after intervention starts) in the prefrail elderlies. | Baseline, 6th, and 12th week of the intervention.
  Handgrip strength will be measured by Hand dynamometer
To assess the changes in dietary intake (Energy, protein) for interventional group (PSG) and control group (CG) from pre-intervention and post-intervention. | Baseline, and 12th week of the intervention.
  Three-day weighed food diaries will be collected at baseline, and postintervention and will be reviewed by the dietitian for completeness. Three-day food diaries will be analyzed using Nutritionist Pro commercial software (version 4.1 Axxya Systems, Stafford TX) to estimate the energy and protein intake (g/kg/day) for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Associate Professor Dr Siti Nur 'Asyura B Adznam, Ass.prof, Principal Investigator — University Putra Malaysia

IPD SHARING:
Plan to Share IPD: No